CLINICAL TRIAL: NCT02737228
Title: A Phase I/II Study of Combination Therapy of CG200745 PPA With Gemcitabine and Erlotinib to Determine the Maximum Tolerated Dose (MTD) and Evaluate the Safety and Efficacy for Locally Advanced Unresectable, or Metastatic Pancreatic Cancer
Brief Title: Study of CG200745 PPA in Combination With Gemcitabine and Erlotinib for Advanced Pancreatic Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CrystalGenomics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CG200745-2-03
Record Dates: First submitted 2016-03-22; First posted 2016-04-13 (Estimated); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — phosphoric acid; Gemcitabine; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CG200745 PPA (Experimental): CG200745 PPA plus Gemcitabine and Erlotinib
  Interventions: Drug: CG200745 PPA; Drug: Gemcitabine; Drug: Erlotinib

INTERVENTIONS:
Drug: CG200745 PPA — CG200745 PPA IV every week three times per cycle (4 weeks)
  Other Names: CG200745 PPA (phosphoric acid)
Drug: Gemcitabine — 1000 mg/m^2 intravenously every week three times per cycle (4 weeks)
  Other Names: combination therapy 1
Drug: Erlotinib — 100 mg per oral daily per cycle (4 weeks)
  Other Names: combination therapy 2

SUMMARY:
<Part I - Phase I trial>

The phase I clinical trial is to identify the MTD (Maximum Tolerated Dose) and DLT (Dose Limiting Toxicity) of CG200745 PPA in combination use of Gemcitabine and Erlotinib. Initial dose of CG200745 PPA is 187.5 mg/m^2, and it will be extended to 250 mg/m^2, 312.5 mg/m^2 or it will be reduced to 125 mg/m^2 based on the results of the cohort of 3 subjects per dose level.

Based on the 3+3 dose escalation study design, Gemcitabine and Erlotinib are administered as fixed doses, whereas CG200745 PPA is to be administered as in four different cohorts according to the dose level. Each cohort consists of 3 or 6 subjects.

<Part II - Phase II trial>

In the phase II clinical trial, the subjects will be administered with the dose which is to be identified as a recommended dose based on the results of Phase I study. The whole one cycle is consisted of 28 days, same as the phase I. The entire treatment period is 6 cycles and tumor assessment is evaluated every 2 cycles.

DETAILED DESCRIPTION:
<Part I - Phase I trial>

The phase I clinical trial is to identify the MTD and DLT of CG200745 PPA in combination use of Gemcitabine and Erlotinib. Initial dose of CG200745 PPA is 187.5 mg/m^2, and it will be extended to 250 mg/m^2, 312.5 mg/m^2 or it will be reduced to 125 mg/m^2 based on the results of the cohort of 3 subjects per dose level.

Based on the 3+3 dose escalation study design, Gemcitabine and Erlotinib are administered as fixed doses, whereas CG200745 PPA is to be administered as in four different cohorts according to the dose level. Each cohort consists of 3 or 6 subjects.

* Dose level 0: CG200745 PPA 125 mg/m^2 puls Gemcitabine 1000 mg/m^2) and Erlotinib 100 mg
* Dose level 1: CG200745 PPA 187.5 mg/m^2 puls Gemcitabine 1000 mg/m^2) and Erlotinib 100 mg
* Dose level 2: CG200745 PPA 250 mg/m^2 puls Gemcitabine 1000 mg/m^2) and Erlotinib 100 mg
* Dose level 3: CG200745 PPA 312.5 mg/m^2 puls Gemcitabine 1000 mg/m^2) and Erlotinib 100 mg

<Part II - Phase II trial>

In the phase II clinical trial, the subjects will be administered with the dose which is to be identified as a recommended dose based on the results of Phase I study. The whole one cycle is consisted of 28 days, same as the phase I. The entire treatment period is 6 cycles and tumor assessment is evaluated every 2 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Ages: ≥ 20 and ≤ 75 years
* Subjects who join voluntarily for participation in the study, sign the consent form and are willing to comply the clinical trial procedure
* Subjects who have diagnosed with unresectable, locally advanced, metastatic, histologically and cytologically confirmed pancreatic adenocarcinoma
* ECOG (Eastern Cooperative Oncology Group) performance status: 0-2
* Estimated life expectancy at the time of enrollment is more than 3 months
* Adequate hematological, renal and hepatic function

  * Absolute neutrophil count (ANC) ≥ 1500/mm3, hemoglobin ≥ 9.0 g/dl (eligible if hemoglobin lab values are adjusted with blood transfusion), platelet ≥ 100,000/mm3
  * Within normal range of serum creatinine or creatinine clearance rate (CCr) ≥ 60 ml/min (using Cockcroft-Gault equation )
  * Subjects who have no abnormal serum electrolyte values (including calcium, magnesium, phosphorous and potassium). However, the supplementation therapy is allowed for normalization of serum electrolytes.

    ※ Normal reference range for Calcium: 8.3~10.5 mg/dl, Magnesium: 1.58~3.0 mg/dl, Phosphorous: 2.4~4.5 mg/dl, Potassium: 3.3~5.5 mmol/L
  * Serum bilirubin < 2 x Upper Limit Normal (ULN), Aspartate Aminotransferase (AST)/Alanine Aminotransferase (ALT) < 2.5 x ULN, Alkaline phosphatase (ALP) < 5 x ULN (If liver metastasis, AST/ALT <5 x ULN)
  * Prothrombin Time (PT) or Partial thromboplastin time (PTT) ≤ 1.5 x ULN (except for the use of anticoagulant, in this case, PT/PTT stabilization for up to 2 weeks should be confirmed)
* No prior chemotherapy, radiation or biologics

Exclusion Criteria:

* Subject who had experienced a major surgery within 2 weeks prior to the screening visit
* Subject with an evidence for uncontrolled brain metastasis (except for the patients with radiologically and neurologically stable brain metastasis without corticosteroid therapy for at least two weeks)
* Subject who cannot be administered oral drug, or have difficulty to absorb the study drugs due to a history of major gastrointestinal surgery or pathological findings.
* Subjects who have treated antibiotics within last seven days due to an active bacterial infection prior to the enrollment. (Topical antibiotic therapies are excluded)
* Subjects who had experienced any malignancies within past 5 years, except for basal cell skin cancer, in situ cervical cancer, or papillary thyroid tumor.
* Pregnancy or Lactating
* Fertile subjects who do not agree with the effective contraception during the study period and up to 3 months after the completion of the study. The following cases are exceptions: an irreversible and surgical sterility by hysterectomy, bilateral oophorectomy or bilateral salpingectomy, and menopausal women over 50 years old with no menstruation for at least 12 months and without hormonal therapy. Tubal ligation is not regarded as an effective contraception
* Subject who cannot take anti-cancer chemotherapy due to a systemic disease (ex. chronic renal failure)
* Subjects who have treated with any other investigational drug within 4 weeks prior to the screening visit
* History of hypersensitivity to study drug
* Subject with HIV positive

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-03; Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | up to 6 cycles (each cycle is 28 days)
  ORR is the proportion of the subjects with CR and PR in comparison to the total subjects at the final tumor assessment point (cycle 6) from the baseline

SECONDARY OUTCOMES:
Disease control rate (DCR) | up to 6 cycles (each cycle is 28 days)
  DCR is the proportion of the subjects with Complete Response (CR), Partial Response (PR), and stable disease (SD) in comparison to the total subjects at the final tumor assessment point (cycle 6) from the baseline
Area Under the Curve [AUC] | before the administration and up to 1440 mins after completion of the IP (Investigational Product) administration
  Pharmacokinetics (PK) parameter
Maximum Plasma Concentration [Cmax] | before the administration and up to 1440 mins after completion of the IP administration
  Pharmacokinetics (PK) parameter
Adverse Events | up to 6 cycles (each cycle is 28 days)
  safety parameter
Clinical laboratory tests | up to 6 cycles (each cycle is 28 days)
  safety parameter

CONTACTS AND LOCATIONS:
Overall Officials: Siyoung Song, M.D., PhD., Principal Investigator — Yonsei University
Locations (1):
- Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided